CLINICAL TRIAL: NCT04203030
Title: Physical Activity to Improve Physical Function in a Community-Based Health Ministry in Chicago's West Side
Brief Title: Physical Activity to Improve Physical Function in a Community-Based Health Ministry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Brittney Lange-Maia, Assistant Professor in Preventive Medicine, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORA18122105
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Aging; Mobility Limitation
Keywords: aging; physical function
MeSH Terms: conditions — Mobility Limitation | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Activity (Experimental): 16 week physical activity intervention
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — Participants will meet in a weekly group session to discuss a topic related to physical activity and physical function and participate in group-based physical activity. Participants will also have instructions to participate in physical activity outside of the weekly sessions, incrementally increasing their total physical activity over the intervention period.

SUMMARY:
This study is being conducted to test if a program with physical activity and learning about movement (including goal setting, benefits of physical activity, and how to increase physical activity gradually) helps people to become more active and to move better. The physical activity program involves specific exercises done in a group setting, and the education part will involve learning about different ways to move to make everyday activities easier. The program will last 16 weeks. This program will take place in a large fellowship area of a partner church through an established community-based participatory research partnership in Chicago, IL.

DETAILED DESCRIPTION:
Limitations in physical function (PF) are related to decreased quality of life and are predictive of disability, nursing home admission, increased healthcare costs, and mortality in older adults. Structured physical activity has been shown to prevent mobility disability among those with physical function limitations, though community-based programs are needed, particularly in underserved communities. The purpose of this study is to pilot test a tailored physical activity intervention in churches in Chicago's West Side through an existing community-based participatory research partnership. The investigators previously found high rates of physical function limitations in these communities, and through qualitative research have identified intervention components that may aid in promoting physical activity among community members with physical function limitations. The primary aim is test the intervention in a 16 week, proof-of-concept study in 20 participants who are ambulatory but have PF limitations. The group-based physical activity intervention will take place in a large common area of a church. For feasibility the investigators will be testing the intervention in one church. The intervention will be delivered over 16 weeks, with assessments at baseline and 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 or older
2. Not currently participating in another formal exercise program and perform less than 150 minutes per week of exercise
3. Ambulatory, defined as able to get out of a chair and walk without assistance aside from using a straight cane.
4. Have any difficulty: Walking ¼ mile, (about 2-3 blocks) OR Walking up 10 steps without resting
5. Speak English
6. Safe to begin an exercise program (determined using the Exercise Assessment and Screening for You (EASY) Tool. Physician clearance may be needed based upon EASY Screening recommendations

Exclusion Criteria:

1. Severe cognitive impairment, defined as five or more errors on the Short-Portable Mental Status Questionnaire
2. Plans to move out of the geographic area during the study period
3. Plans to have major surgery within the study period Anticipate having major schedule changes that would interfere with ability to participate in the program.
4. Inability to get to intervention location on a weekly basis
5. Unwilling to commit to a weekly, approximately 90 minute program for 16 weeks.
6. Contraindications to exercise determined using the EASY/healthcare follow-up.
7. Self-reported

   * Heart disease
   * Uncontrolled diabetes mellitus
   * Pacemaker
   * Stroke within past 12 months
   * Severe chronic lung disease (emphysema or COPD)
   * Recent healing or unhealed fractures in the past 6 months
   * Heart failure
   * Chronic kidney disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Physical Function | 16 weeks
  Change in Short Physical Performance Battery score Scale ranges from 0-12 (integers only) with higher scores indicating better function.

SECONDARY OUTCOMES:
Physical Activity (Objective) | 16 weeks
  Change in accelerometer measured physical activity (minutes of moderate/vigorous physical activity per day, and number of steps per day). Accelerometer will be worn for 1 full week at the hip but removed for sleep at night). Higher positive values of change indicate larger increases in physical activity.
Physical Activity (Self-Reported) | 16 weeks
  Change in physical activity as assessed by the Champs physical activity. questionnaire. Activity will be expressed as caloric expenditure/week in all exercise-related activities (in calories per week). Higher positive values of change indicate larger increases in physical activity.
Acceptability of intervention: | 16 weeks
  Acceptability questionnaire specific to intervention, attendance (% of sessions attended out of 16 total)

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No